CLINICAL TRIAL: NCT06348069
Title: Pharmacy-based PrEP for Young Women Who Sell Sex in Zimbabwe
Acronym: TOPAZ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Centre for Sexual Health and HIV/AIDS Research Zimbabwe (CeSHHAR Zimbabwe) (Other); University of California, San Francisco (Other); Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-11-15783
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Adherence, Medication; HIV Prevention
Keywords: HIV; PrEP; People who engage in sex work
MeSH Terms: conditions — Medication Adherence | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Groups (sites/clusters) are randomized to either the intervention (pharmacy-based PrEP refills plus gift card incentives) or the control (standard of care) and are followed and compared over time.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacy-based PrEP refills + gift cards (Experimental): Participants who have, in addition to the standard practice of refill pickups at CESHHAR clinics, the opportunity to retrieve PrEP refills at private pharmacies, and who receive gift card incentives at the designated refill time-points of 1, 3, and 6 months.
  Interventions: Behavioral: Pharmacy-based PrEP refill and gift voucher
- Control (Standard of Care) (Experimental): Participants who do not have the opportunity to retrieve PrEP refills at private pharmacies. PrEP refill pick-ups are available through CESHHAR Zimbabwe's existing network of clinical sites.
  Interventions: Behavioral: Control (Standard of care)

INTERVENTIONS:
Behavioral: Pharmacy-based PrEP refill and gift voucher — The intervention arm of this study introduces the opportunity for a pharmacy-based PrEP refill system for sex workers, coupled with financial incentives to increase adherence. Participants receive PrEP medications from selected pharmacies, a strategy designed to improve PrEP access and enhance privacy/discretion. Additionally, participants in the intervention are awarded escalating gift card values for each successful refill collection at study pharmacies, aiming to incentivize continued PrEP use for effective HIV prevention. The intervention seeks to enhance convenience and motivate adherence through financial rewards.
  Arms: Pharmacy-based PrEP refills + gift cards
Behavioral: Control (Standard of care) — For sex workers in the control group, PrEP refill pick-up will be available through CESHHAR's existing network of clinical sites. There is no gift card incentive and no pick-up at private pharmacies.
  Arms: Control (Standard of Care)

SUMMARY:
Pharmacy-based PrEP for Young Women who Sell Sex in Zimbabwe is a cluster-randomized control trial and pilot study co-led by Dr. Euphemia Sibanda, Reader (Associate Professor) of Global Health and Epidemiology at Liverpool School of Tropical Medicine, UK and Research Director at the Centre for Sexual Health and HIV Research (CeSHHAR Zimbabwe) and Dr. Sandra McCoy, Professor of Epidemiology and Biostatistics at the University of California, Berkeley. The goal of the proposed study is to optimize, refine and pilot a pharmacy-based PrEP intervention for female sex workers (FSW) in Zimbabwe. Despite efforts to reach the most impacted and vulnerable populations with PrEP, retention rates, particularly among FSW in Africa, are very low. Relatively high levels of uptake indicate that FSW are interested in PrEP and ready to initiate it, but in most cases fewer than 50% of those who initiate return for medication refills by month 4. Pharmacy-based PrEP has the potential to address known barriers to PrEP retention among FSW such as stigma and access, and coupled with a small escalating incentive in the form of a gift card incentive, could also boost motivation for effective use of PrEP.

ELIGIBILITY:
Inclusion Criteria:

* 1) Exchanged sexual intercourse for money or gifts in past 6 months
* 2) Age 16 or older
* 3) HIV negative (via rapid test per national guidelines) at enrollment and no signs/symptoms of acute HIV infection

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-03-11 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PrEP retention at 6 months | 6 months
  This will be measured as attendance within one week (before and after) of the scheduled refill visit at the 6-month visit. Outcome 1 will also be measured as follows: Proportion of visits completed as scheduled, by arm.

OTHER OUTCOMES:
PrEP retention at 6 months among FSW who are 18-24 years of age | 6 months
  : PrEP retention at 6 months among FSW who are 18-24 years of age, stratified by pickup location. This will be measured as attendance within one week (before and after) of the scheduled refill visit at the 6-month visit. Outcome 2 will also be measured as follows: Proportion of visits completed as scheduled, by arm.
: PrEP retention at 6 months among participants who have remained active in sex work | 6 months
  PrEP retention at 6 months among participants who have remained active in sex work (based on program, referral app and microplanner data). This will be measured as attendance within one week (before and after) of the scheduled refill visit at the 6-month visit. Outcome 3 will also be measured as follows: Proportion of visits completed as scheduled, by arm.
FSW (overall) and FSW (18-24 years) patronage for PrEP services at pharmacies | 9 months
  FSW (overall) and FSW (18-24 years) patronage for PrEP services at pharmacies, defined as the proportion of PrEP refill pick-ups in intervention suburbs occurring at pharmacies.
HIV tests | 9 months
  The number and outcomes of HIV tests at the time of refill.
HIV care referrals | 9 months
  This outcome will measure the number of referrals for HIV care.

CONTACTS AND LOCATIONS:
Locations (1):
- CESHHAR Zimbabwe, Harare, Zimbabwe

REFERENCES:
- [Derived] Kuguyo O, Archer H, Azizi L, Watadzaushe C, Munhenzva S, Chidhanguro K, Takaruza A, Musemburi S, Packel L, Liu J, Matambanadzo P, Cowan FM, McCoy S, Sibanda EL. Establishing a Pharmacy-Based Pre-Exposure Prophylaxis Program for Young Women Who Sell Sex: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Dec 3;14:e74141. doi: 10.2196/74141. PMID 41337741